CLINICAL TRIAL: NCT03854929
Title: An Open Label Randomised Controlled Trial of Azithromycin Versus Ciprofloxacin for the Treatment of Children Hospitalised With Dysentery in Ho Chi Minh City, Vietnam
Brief Title: Ciprofloxacin Versus Azithromycin for Children Hospitalised With Dysentery
Acronym: CIPAZ
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Oxford University Clinical Research Unit, Vietnam (Other)
Collaborators: Number 2 Children's Hospital, Ho Chi Minh City (Other); University of Liverpool (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 26EN
Record Dates: First submitted 2019-02-21; First posted 2019-02-26 (Actual); Last update posted 2023-06-07 (Actual); Status verified 2023-06

CONDITIONS: Dysentery, Shigella; Shigellosis; Diarrhea
Keywords: Azithromycin; Ciprofloxacin; Children; Dysentery; Vietnam
MeSH Terms: conditions — Dysentery, Bacillary; Diarrhea; Dysentery | interventions — Ciprofloxacin; Azithromycin

STUDY DESIGN:
Intervention Model Description: Randomization will be 1:1 to either AZI or CIP. Block randomization with stratification by hospital of enrolment, and variable block sizes of 4 and 6, respectively, will be used to assign subjects to treatment. The randomization list will be generated according to standard operating procedures without our organization. In brief, the Research Biostatistician (RB) will generate a randomization list using an in-house statistical code and transfer it to the central Study Pharmacist (SP). The SP will change the random seed to blind the RB and then run the code to prepare the final randomization list for treatment preparation. The randomization list will be saved and stored on a secure server.
  After enrolment, children will be randomly allocated to one of two treatment arms: in one arm, children will be treated with the current standard of care, oral CIP 15mg/kg BW /twice daily for 3 days, while those in the other arm will receive oral AZI 10mg/kg BW/daily for 3 days.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ciprofloxacin (Active Comparator): Each sachet CIPROFLOXACIN of 3g powder contains: 250mg Ciprofloxacin HCl, dissolved in water, dosed to 15mg/kg body weight /twice daily (apart 12 hours)/ 3 days.
  Interventions: Drug: Ciprofloxacin
- Azithromycin (Experimental): Each sachet AZICINE of 1.5 g powder contains: 250mg of Azithromycin dihydrate, dissolved in warm water, dosed to 10mg/kg body weight /daily/ 3 days
  Interventions: Drug: Azithromycin

INTERVENTIONS:
Drug: Ciprofloxacin — Fluoroquinolone, ATC code: J01MA02
  DNA-gyrase and topoisomerase IV inhibitor
  Arms: Ciprofloxacin
Drug: Azithromycin — Macrolide, ATC code: J01FA10
  Binds to ribosomal 50S sub-unit inhibiting translocation of peptides thereby suppressing bacterial protein synthesis.
  Arms: Azithromycin

SUMMARY:
The purpose of this study is to assess the efficacy of 3 days of azithromycin (AZI) compared to 3 days of ciprofloxacin (CIP) (standard-of-care) for the treatment of children hospitalised with dysentery in Ho Chi Minh City.

DETAILED DESCRIPTION:
Antimicrobial resistance is a well-established international healthcare crisis and children with diarrhoeal infections represent a significant proportion of the global infectious disease burden. With the increasing rates of antimicrobial resistance observed in the organisms associated with children presenting with dysentery in Vietnam and the investigator's capacity to demonstrate international transmission events, new data regarding alternative treatment options such as azithromycin, in particular for the new highly-antimicrobial resistant S. sonnei, are urgently needed.

The study team will perform a phase IV open label randomised controlled trial to compare the efficacy of AZI to CIP (standard-of-care) for the treatment of children hospitalised with dysentery in Ho Chi Minh City, Vietnam. Children aged 6 to 60 months presenting to the participating hospital with symptoms/signs of dysentery (diarrhoea with blood and/or mucus accompanied by 1 or more of: fever ≥37.8°C, abdominal pain and /or tenesmus) within the previous 72 hours will be enrolled to the study.

After enrolment, participants will be managed according to WHO and local algorithms for children with bloody diarrhoea. In addition, after providing a stool sample, children will be randomly allocated to receive CIP 15mg/kg body weight/ twice daily or AZI 10mg/kg body weight/ daily for 3 days. After enrolment, children will be reviewed for clinical and microbiological response to treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female aged 6 months to 60 months at time of hospital presentation.
2. Have symptoms and/or signs of dysentery, specifically passing stools containing mucus and/or blood with/without abdominal pain, tenesmus or fever (≥37.8˚C).
3. Be eligible for treatment with oral medication in the opinion of the admitting physician (i.e. no clinical requirement for parenteral treatment on admission).
4. Be within 72 hours of the onset of signs/symptoms.
5. Have a parent/guardian present at admission who can provide written informed consent.

Exclusion Criteria:

1. Those known to have specific medical (patients with known prolongation of the QT interval, congenital long QT syndrome)/surgical conditions which may affect disease severity/presentation or response to treatment (e.g. affecting antimicrobial absorption), including:

   1. gastrointestinal abnormalities, including short bowel syndrome, chronic (inflammatory or irritable) bowel disease.
   2. inherited or acquired immune system deficiency rendering the patient immunocompromised, including chronic/long-term steroid treatment or other immunosuppressive treatment
2. Presentation with severe infection requiring parenteral antimicrobial treatment, including shock jaundice, extensive gastrointestinal bleeding, convulsion , drowsiness or coma, reduced or less movement when stimulated, tachypnea > 60 times per minute, grunting, chest retraction, refuse to suck.
3. Known hypersensitivity to any of the trial drugs (CIP or AZI).
4. Coexisting infection requiring other or additional antimicrobials to be prescribed/ administered.

Ages: 6 Months to 60 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 364 (Actual)
Dates: Start 2019-12-11 (Actual); Primary Completion 2021-02-06 (Actual); Study Completion 2022-07-12 (Actual)

PRIMARY OUTCOMES:
Assess the Clinical treatment failure between treatment groups. | after 120 hours of start of either treatment.
  Clinical treatment failure including: fever ≥38.0°C or the persistence of signs or symptoms of the infection (vomiting, abdominal pain, passing loose stools more than 3 times per 24 hours ( with blood and mucus, blood or mucus, without both))
Assess the microbiological treatment failure between treatment groups. | after 72 hours of start of either treatment.
  The microbiological treatment failure is assessed by positive PCR stool with original pathogen after day 3 of treatment.

SECONDARY OUTCOMES:
Measure differences in symptom duration between treatment groups by stratifying stool PCR. | 120 hours of start of either treatment.
  Compare the duration of symptom ( from the onset to disappear) between the two groups.
  The duration of symptom will be stratified by stool PCR.
Measure differences in symptom duration between treatment groups by stratifying stool culture. | 120 hours of start of either treatment.
  Compare the duration of symptom ( from the onset to disappear) between the two groups.
  The duration of symptom will be stratified by stool culture.
Assess the time to resolution of objective markers of infection and inflammation, including cessation of culture- and PCR-confirmed Shigella shedding, normalization of blood total white cell count, C-reactive protein and stool lipocalin | at enrolment, day 7th (+3 days) and day 28th (+3 days)
  Time to cessation of Shigella shedding in stool (PCR).
Assess the rates of adverse events associated with exposure to the antimicrobial agents used. | at enrolment, during 31 days after enrolment
  Adverse effects of antimicrobial treatment, including (i) life-threatening events, (ii) events requiring drug discontinuation, (iii) mild adverse events that require additional medication to be used but not resulting in drug discontinuation.
Assess the effects of antimicrobial exposure on the host microbiome, including diversity and abundance of specific bacterial species in stool. | at enrolment, day 7th (+3 days) and day 28th (+3 days).
  The extend of intestinal microbial colonisation will be assessed by analyses of stool sample collected at enrolment, day 7th (+3 days) and day 28th (+3 days)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Stephen, Professor, Principal Investigator — Oxford University Clinical Research Unit
Locations (1):
- Children's Hospital 2, Ho Chi Minh City, Vietnam

IPD SHARING:
Plan to Share IPD: Undecided